CLINICAL TRIAL: NCT07293949
Title: Ultrasonographic Evaluation of Talar Cartilage Thickness in Patients With Spinal Cord Injury: A Cross-Sectional Case-Control Study
Brief Title: Ultrasonographic Evaluation of Talar Cartilage Thickness in Patients With Spinal Cord Injury
Status: Recruiting | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 172
Record Dates: First submitted 2025-11-22; First posted 2025-12-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries (SCI); Osteoarthritis (OA)
Keywords: spinal cord injury; osteoarthritis; musculoskeletal ultrasound; talar cartilage
MeSH Terms: conditions — Spinal Cord Injuries; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: Spinal cord injury patients
- Control group: Age, sex, and BMI matched healthy controls

SUMMARY:
Spinal cord injury patients often present with musculoskeletal comorbidities, including osteoarthritis. Early detection of cartilage damage is important for preventing osteoarthritis progression. This study aims to compare the talar cartilage thicknesses of spinal cord injury patients with healthy subjects. The secondary aim is to investigate a correlation between the talar cartilage thickness and disease-related parameters. The patient group is to be assessed for talar cartilage thickness (via ultrasound), functional status, spasticity, and ambulation levels.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 to 60 years,
* Cervical, thoracal or lumber level of spinal cord injury
* AIS (American Spinal Injury Association Impairment Scale) Level A, B, C, or D
* Assisted ambulation of any kind
* Literacy
* Giving oral and written consent to participate in the study

Exclusion Criteria:

* Patients with sacral level injury
* AIS E
* MAS 4 level of spasticity
* History of any lower extremity operation
* History of fracture
* Botulinum toxin injection in the last 6 months
* Existing diagnosis of any rheumatologic or endocrine diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thirty-eight SCI patients who apply to Physical Medicine and Rehabilitation outpatient and inpatient clinic between November 2025-January 2026 will be included in the study.
  Thirty-eight age, gender, and BMI-matched healthy participants who are literate, give oral and written consent without any additional disease will be formed as the control group.
Sampling Method: Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Talar cartilage thickness | Baseline
  The talar cartilage of both lower extremities are to be assessed with ultrasound

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) score | Baseline
  Functional Independence Measure scores will be held for the patient group in order to assess functional independence. This 18-item scale ranges between 18-126, higher scores indicating better outcomes.
Modified Ashworth Scale (MAS) | Baseline
  The spasticity level of patients are to be recorded for both ankle flexor and extensors via Modified Ashworth Scale. This scale ranges from 0 to 4; 0 indicating no spasticity, and 4 indicating severe increase in muscle tone with rigid joint.
Walking Index for Spinal Cord Injury II (WISCI II) | Baseline
  Ambulatory status of the patients will be recorded with this measuring scale, ranging between 0 (non ambulatory) to 20 (able to walk 10 meters with no devices/orthosis/assistance).

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The datasets of the study (patient and volunteer demographics, clinical data, and statistical data) will be shared after completion of the study with third parties upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 3 years after the publication of results